CLINICAL TRIAL: NCT07192263
Title: A Phase 3, Multi-center, Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate the Efficacy and Safety of IN-B00009 Injection in Adults With Obesity or Overweight Without Diabetes Mellitus
Brief Title: Study to Evaluate the Efficacy and Safety of IN-B00009 Injection in Adults With Obesity or Overweight Without Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN_ECN_301
Record Dates: First submitted 2025-09-08; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Obesity &Amp; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IN-B00009 (Experimental)
  Interventions: Drug: IN-B00009
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IN-B00009 — Test drug
  Arms: IN-B00009
Drug: Placebo — Placebo drug
  Arms: Placebo

SUMMARY:
This Phase 3 study is designed to evaluate the efficacy and safety of IN-B00009 injection in adults with obesity or overweight without diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 to 75 years as of the date of written consent
2. Those who meet any of the following obesity criteria at the screening visit

   * BMI ≥ 30 kg/m2
   * 27 kg/m2 ≤ BMI < 30 kg/m2 with at least one risk factor or comorbidity

     * BMI (kg/m2) = weight (kg) / height (m)2

       * Hypertension: Taking antihypertensive medication or sitSBP ≥ 140 mmHg or sitDBP ≥ 90 mmHg
       * Dyslipidemia: Taking dyslipidemia medication or Total Cholesterol ≥ 240mg/dL or LDL-C ≥ 160 mg/dL or TG ≥ 200 mg/dL or HDL-C < 40 mg/dL
       * Obstructive sleep apnea
       * Cardiovascular and cerebrovascular diseases: Ischemic cardiovascular and cerebrovascular diseases not corresponding to exclusion criterion 17, heart failure of NYHA Class I to III, etc.
       * Prediabetes: 100 mg/dL ≤ FPG ≤ 125 mg/dL or 140 mg/dL ≤ PG ≤ 199 mg/dL at 2 hours after 75 g oral glucose load or 5.7% ≤ HbA1c ≤ 6.4%
3. Self-reported history of at least one failed attempt at weight control using diet and exercise therapy prior to the screening visit
4. Able to agree to and follow the reduced-calorie diet and exercise therapy recommended in this study during the study period
5. Agrees to use a medically appropriate method of contraception (including medically infertile conditions) during the study period

Exclusion Criteria:

1. Body weight change exceeding 5 kg within 3 months of the screening visit
2. Diabetes (Type 1, Type 2, etc.) or HbA1c ≥ 6.5% at the screening visit
3. Received any of the following medications or treatments within 3 months of the screening visit

   ① Obesity-related medications (such as GLP-1 receptor agonists) or medications including over-the-counter drugs, herbal medicines, or health functional foods for weight control

   ② Received hypoglycemic agent or requires continuous administration during the study period

   ③ Received systemic steroids for 30 consecutive days or more, or requires continuous administration during the study period

   ④ Received other medications that cause significant body weight changes or requires continuous administration during the study period (e.g.: antipsychotics, tricyclic antidepressants, selective serotonin reuptake inhibitors, noradrenergic and specific serotonergic antidepressant, mood stabilizers (lithium), anticonvulsants, serotonin antagonists, first-generation antihistamines, etc.)
4. Diagnosed with obesity due to endocrine disorders (hypothalamic obesity, Cushing's syndrome, insulinoma, adult growth hormone deficiency, hypothyroidism, etc.)
5. Diagnosed with obesity due to genetic variations and congenital disorders

   * Obesity-causing genes: ob, db, Proopiomelanocortin (POMC), Melanocortin 4 receptor (MC4R) genes, etc.
   * Congenital disorders: Prader-Willi syndrome, Laurence-Moon-Biedl syndrome, Alström syndrome, Cohen syndrome, Carpenter syndrome, etc.
6. History of bariatric surgery (e.g., adjustable gastric banding, sleeve gastrectomy, Roux-en-Y gastric bypass, biliopancreatic diversion/duodenal switch, etc.) or device procedures, or plans for such during the study period

   * However, those who have had devices (e.g., gastric band, intragastric balloon) removed for more than 1 year can participate
   * Those who have had liposuction or abdominoplasty for more than 1 year can participate
7. Clinically significant gastrointestinal disorders (e.g., gastroparesis, gastric outlet obstruction, peptic ulcer, severe gastroesophageal reflux disease)
8. History (including family history) of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2), or results of clinical laboratory test at the screening visit meeting the following:

   * Calcitonin ≥ 100 ng/L
   * TSH < 0.6 mIU/L or TSH > 6.8 mIU/L (However, subjects being treated for hypothyroidism with 0.6 mIU/L ≤ TSH ≤ 6.8 mIU/L, taking stable doses of thyroid hormonal preparation for 3 months prior to the screening visit and unlikely to have dose changes during the study period can participate)
9. History of acute or chronic pancreatitis, or results of clinical laboratory test at the screening visit meeting the following:

   - Amylase or Lipase > 3 times the upper limit of normal
10. Severe hepatic impairment or results of clinical laboratory test at the screening visit meeting the following:

    - AST or ALT > 3 times the upper limit of normal or Total bilirubin > 2 times the upper limit of normal
11. Severe renal impairment (eGFR < 30mL/min/1.73m2)
12. Uncontrolled hypertension (sitSBP ≥ 160 mmHg or sitDBP ≥ 100 mmHg) at the screening visit
13. Answered "yes" to question 4 or 5 in the suicidal ideation section of the Columbia-Suicide Severity Rating Scale (C-SSRS) at the screening visit or history of suicide attempt
14. Score of 15 or higher on the Patient Health Questionnaire-9 (PHQ-9) at the screening visit, or history of major depressive disorder with unstable state, anxiety, or other severe psychiatric disorders (schizophrenia, bipolar disorder, etc.) within 2 years
15. History of alcohol addiction or drug abuse within 3 months of the screening visit
16. History of malignant tumor within the last 5 years

    * Those who have been determined as complete remission (CR, pCR) of the tumor and had no relapse for 5 years or more from the date of assessment can participate
    * Those with a history of thyroid cancer (excluding MTC), basal cell and squamous cell skin cancer within the last 5 years can participate
17. Any of the following medical histories confirmed within 3 months of the screening visit

    * Heart failure of NYHA class IV
    * Coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI)
    * Ischemic heart disease (acute myocardial infarction, unstable angina, etc.). However, if the condition has been stable for 6 months or more from the screening visit, participation is possible at the investigator's discretion
    * Severe cerebrovascular disease (cerebral infarction, cerebral hemorrhage, etc.), transient ischemic attack (TIA). However, if the condition has been stable for 6 months or more from the screening visit, participation is possible at the investigator's discretion
18. History of non-arteritic anterior ischemic optic neuropathy (NAION)
19. History of resistance or hypersensitivity to investigational product class drugs (GLP analogues) or history of multi-drug allergies
20. Requires administration of contraindicated medications during the study period
21. Received other investigational products within 30 days or 5 times the half-life (whichever is longer) if the half-life is known, prior to the screening visit
22. Positive for HBsAg, HCV antibody, or HIV antibody at the screening visit

    - However, those who are HCV-Ab positive but confirmed negative in HCV-RNA test can participate
23. Hematological conditions that may interfere with HbA1c measurement (e.g.: hemolytic anemia, hemoglobinopathies)
24. Scheduled for surgery requiring hospitalization during the study period or requires surgical treatment
25. Positive pregnancy test, pregnant or lactating women
26. Considered inappropriate as a study subject by the investigator for other reasons

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in body weight from baseline at Week 40 | Baseline, 40 weeks
Proportion of subjects with ≥5% body weight loss from baseline at Week 40 | Baseline, 40 weeks

SECONDARY OUTCOMES:
Percent change in body weight from baseline at Week 24 | Baseline, 24 weeks
Proportion of subjects with ≥5% body weight loss from baseline at Week 24 | Baseline, 24 weeks
Proportion of subjects with ≥10% body weight loss from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks
Proportion of subjects with ≥15% body weight loss from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks
Change in body weight from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks
Change in BMI from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks
Change in waist circumference from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks
Change in glucose metabolism parameters from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks
Percent change in lipids from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks
Change in blood pressure(systolic, diastolic) from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks
Change in IWQOL-Lite-CT(Impact of Weight on Quality of Life-Lite for Clinical Trials version) (Physical function domain) from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks
Change in SF-36(36-Item Short Form Survey) scores from baseline at Week 24 and Week 40 | Baseline, 24 weeks, 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cheol-Young Park, Principal Investigator — Kangbuk Samsung Hospital

IPD SHARING:
Plan to Share IPD: No